CLINICAL TRIAL: NCT00256282
Title: A Phase II Evaluation of Docetaxel and Vinorelbine Plus Sargramostim in Patients With Metastatic Malignant Melanoma
Brief Title: Docetaxel and Vinorelbine Plus Sargramostim in Metastatic Malignant Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John P. Fruehauf (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor-Investigator, John P. Fruehauf, Professor of Clinical Medicine, University of California, Irvine
Organization: University of California, Irvine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 02-23; 2002-2763 (Other: University of California, Irvine); NCI-2010-00217 (Other: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Results first posted 2018-05-03 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-02

CONDITIONS: Metastatic Melanoma
Keywords: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Vinorelbine; Docetaxel; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel & Vinorelbine + Sargramostim (Experimental): Docetaxel, Vinorelbine, and Sargramostim
  Interventions: Drug: Vinorelbine; Drug: Docetaxel; Drug: Sargramostim

INTERVENTIONS:
Drug: Vinorelbine — 30 mg/m2 IV over 6-10 min every 14 days
  Other Names: Navelbine; NSC-608210
Drug: Docetaxel — 40mg/m2 IV over 1 hour every 14 days
  Other Names: Taxotere; RP56976; NSC-628503
Drug: Sargramostim — 250 mcg/m2 subcutaneous (SQ) daily (QD) x 10 days
  Other Names: Recombinant GM-CSF; Leukine; Immunex; NSC-613795

SUMMARY:
This is a Phase II Evaluation of Docetaxel and Vinorelbine Plus Sargramostim in subjects who have metastatic melanoma which has advanced beyond the point at which local therapies such as surgery or radiation therapy would be helpful. Without effective treatment, metastatic melanoma is usually a severe and fatal disease. Chemotherapy agents or combinations of chemotherapy agents have produced tumor shrinkage in some patients, which has occasionally persisted. This research involves treatment with a combination of chemotherapy drugs known to be active against melanoma alone. The investigational purpose of this study is to determine if the combination of docetaxel, vinorelbine and sargramostim will produce a response (complete or partial) in metastasis melanoma. The researchers also wants to find out what side effects are associated with this combination of drugs.

DETAILED DESCRIPTION:
Annually in the U.S. there is an estimated 40,000 new cases of malignant melanoma and 7000 deaths. This disease is becoming more common with its incidence increasing at a more rapid rate in the past decade than that of any other cancer except lung cancer in women. Metastatic disease responds poorly to the usual treatments with only 2 out of 30 drugs tested, DTIC and nitrosoureas, showing response rates greater than 10%. Complete responses are rare.

Metastatic melanoma is a disease with few therapeutic options. Multi-agent chemotherapy with cisplatin (CDDP), Dacarbazine (DTIC), Carmustine (BCNU), with or without Tamoxifen, offers a 20% response rate but has failed to consistently demonstrate a significant improvement in overall survival (OS) or disease-free survival (DFS) when compared to a single agent DTIC.

Recently, investigators, in an effort to combine the activity of biologic response modifiers with chemotherapy, have developed combination biochemotherapy for metastatic melanoma. Legha et al reported an overall objective response rate of 64% with a 5-day biochemotherapy regimen. O'Day et al reported similar results (overall response rate of 57%) using a modified 5-day biochemotherapy regimen.

The above regimens all have significant toxicities and modest response rates. Clearly, more effective less toxic regimens are needed.

Vinorelbine tartrate (Navelbine) and Docetaxel (Taxotere) have both shown activity against melanoma. Additionally, the combination of both drugs has shown enhanced activity against melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18
* Karnofsky Performance Status (KFS) of greater than or equal to 70
* Laboratory values (performed in 14 days, inclusive prior to study drug administration):

  * Absolute neutrophil count (ANC) >1500/mm3
  * Platelet count >100,000/mm3
  * Hemoglobin > 10 g/dl
  * Blood urea nitrogen (BUN) and serum creatinine < 0.5 times the upper limit of laboratory normal
  * Total and direct bilirubin < 1.5 times the upper limit of laboratory normal
  * Serum glutamic-oxaloacetic transaminase (SGOT) and Serum glutamic pyruvic transaminase(SGPT) < 3 times the upper limit of laboratory normal
  * Alkaline phosphatase < 3 times upper limit of laboratory normal
* Life expectancy of greater than 12 weeks
* Written informed consent

Exclusion Criteria:

* No recovery from all active toxicities of prior therapies
* Surgery within 1 week prior to study drug administration, providing acute surgical toxicity is resolved
* Subjects within acute infection treated with intravenous antibiotics
* Frequent vomiting or medical condition that could interfere with oral medication intake (e.g., partial bowel obstruction)
* Concurrent malignancies at other sites with the exception of surgically cured carcinoma in situ (CIS ) of the cervix, basal or squamous cell carcinoma of the skin, and prior malignancies which have not required anit-tumor treatment within the preceding 24 months
* Known HIV-positivity or AIDS-related illness
* Women of childbearing potential who are not using an effective method of contraception (eligible patients must have a negative urine pregnancy test 24 hours prior to administration of study drug and be practicing medically approved contraceptive precautions)
* Men who do not use an effective method of contraception.
* Chemotherapy within four weeks prior to study drug administration or biologic therapy/immunotherapy within two weeks prior to study drug administration
* Completion of radiation therapy, interstitial brachytherapy, or radiosurgery within 4 weeks prior to study drug administration (patients with brain metastases from melanoma must have completed radiotherapy to the brain at least 3 weeks before study commences)
* Bone metastases as sole reason for Stage IV disease
* Karnofsky Performance Status of less than or equal to 60

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P. Fruehauf, MD, PhD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eroglu Z, Kong KM, Jakowatz JG, Samlowski W, Fruehauf JP. Phase II clinical trial evaluating docetaxel, vinorelbine and GM-CSF in stage IV melanoma. Cancer Chemother Pharmacol. 2011 Oct;68(4):1081-7. doi: 10.1007/s00280-011-1703-z. Epub 2011 Jul 19. PMID 21769667

RESULTS

PARTICIPANT FLOW:
Groups:
- Docetaxel and Vinorelbine Plus Sargramostim: Docetaxel (40 mg.m2 IV), Vinorelbine (30 mg/m2 IV), and Sargramostim 250 mcg/m2 subcutaneous (SQ)
  Vinorelbine: 30 mg/m2 IV over 6-10 min every 14 days
  Docetaxel: 40mg/m2 IV over 1 hour every 14 days
  Sargramostim: 250 mcg/m2 subcutaneous (SQ) daily (QD) x 10 days
Period: Overall Study
Arm/Group | Docetaxel and Vinorelbine Plus Sargramostim
Started | 52
Completed | 36
Not Completed | 16
Not completed — Disease progression, relapse during acti | 12
Not completed — Adverse Event | 3
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Docetaxel and Vinorelbine Plus Sargramostim: The DVS regimen consisted of docetaxel 40 mg/m2 IV over 1 hour, vinorelbine 30 mg/m2 IV over 6 to 10 minutes on day 1, every 14 days, and GM-CSF, 250 mg/m2 SC on days 2 to 12. Patients received a cycle of this regimen every two weeks.
Arm/Group | Docetaxel and Vinorelbine Plus Sargramostim
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 18
Age, Continuous [Median (Full Range); unit: years] | 62.0 [24 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 36
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) in Patients With AJCC Stage IV Metastatic Melanoma Treated With Docetaxel and Vinorelbine as First-line or Post-first Line (Salvage) Systemic Therapy
Description: The primary endpoint is to evaluate the six-month progression-free survival (PFS) in patients with AJCC stage IV metastatic melanoma treated with docetaxel and vinorelbine as first-line or post-first line (salvage) systemic therapy. Progressive disease is defined as any new lesion or a greater than or equal to 20% increase in the largest perpendicular diameter of the sum of the T-lesions identified on contrast enhanced CT or MRI scan.
Time Frame: Six months from initial treatment
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Docetaxel and Vinorelbine Plus Sargramostim
Number analyzed (Participants) | 52
days | 134 [91 to 214]

2. Secondary Outcome: Percentage of Patients Alive at One Year
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel and Vinorelbine Plus Sargramostim
Number analyzed (Participants) | 52
Participants | 25

ADVERSE EVENTS:
Time Frame: 6 years, 6 months
Arm/Group | Docetaxel and Vinorelbine Plus Sargramostim
All-Cause Mortality (participants affected / at risk) | 15/52
Serious Adverse Events (participants affected / at risk) | 6/52
Other Adverse Events (participants affected / at risk) | 42/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel and Vinorelbine Plus Sargramostim (N=52)
febrile neutropenia (General disorders) | 6 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel and Vinorelbine Plus Sargramostim (N=52)
anemia (Blood and lymphatic system disorders) | 42 (42)
neutropenia (Blood and lymphatic system disorders) | 19 (19)
thrombocytopenia (Blood and lymphatic system disorders) | 9 (9)
neuropathy (Nervous system disorders) | 16 (16)
alopecia (General disorders) | 40 (50)
Injection site reaction (General disorders) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No